CLINICAL TRIAL: NCT00044798
Title: Vascular Depression and Magnetic Stimulation Therapy
Brief Title: Magnetic Stimulation Therapy for Treating Vascular Depression
Acronym: rtms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Robert G. Robinson, MD, UIHC/Psychiatry
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01MH063405 (NIH); R01MH063405 (NIH); DATR A4-GPX
Record Dates: First submitted 2002-09-04; First posted 2002-09-06 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Depressive Disorder; Depression
Keywords: Aged
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Transcranial Magnetic Stimulation; Citalopram

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive treatment with repetitive transcranial magnetic stimulation and citalopram.
  Interventions: Procedure: Repetitive transcranial magnetic stimulation (rTMS); Drug: Citalopram
- 2 (Active Comparator): Participants will receive treatment with sham repetitive transcranial magnetic stimulation and citalopram.
  Interventions: Drug: Citalopram; Procedure: Sham rTMS

INTERVENTIONS:
Procedure: Repetitive transcranial magnetic stimulation (rTMS) — Participants will receive 15 treatments of rTMS over 3 weeks.
  Arms: 1
Drug: Citalopram — After completing treatment with rTMS or sham rTMS, participants will take citalopram for 9 weeks.
Procedure: Sham rTMS — Participants will receive 15 treatments of sham rTMS over 3 weeks.
  Arms: 2

SUMMARY:
This 12-week study will evaluate the effectiveness of repetitive transcranial magnetic stimulation (rTMS) of the brain, followed by citalopram (Celexa®), for treatment of depression associated with small vascular lesions in the brain (vascular depression).

DETAILED DESCRIPTION:
Vascular depression is a condition that typically affects the elderly and is associated with small vascular lesions. It is more resistant to treatment and has a poorer outcome than nonvascular depression. By altering excitability in the cortical area of the brain, rTMS may be an effective treatment neuropsychiatric conditions, particularly depression.

Participants in this study will be randomly assigned to 15 treatments of either rTMS or sham rTMS for 3 weeks. Following treatment, participants will receive citalopram for 9 weeks. Response rates to treatment; relapse rates; the size, number, and location of the vascular lesions; and the amount of regional brain atrophy will be measured. Improvements in activities of daily living, quality of life, and cognitive function will also be also measured.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of unipolar major or minor depressive disorder
* Hamilton Depression Rating Scale score of at least 18
* Depression that is associated with cerebrovascular disease
* Failed at least 1 treatment for vascular depression

Ages: 51 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2001-09; Primary Completion 2007-03 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Response rates to treatment; relapse rates; the size, number, and location of the vascular lesions; and the amount of regional brain atrophy | Measured at Week 12

SECONDARY OUTCOMES:
Improvements in activities of daily living, quality of life, and cognitive function | Measured at Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Health Care, Iowa City, Iowa, United States